CLINICAL TRIAL: NCT02465879
Title: Allied Health in Rheumatology Triage Project
Acronym: AHRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Arthritis Society, Canada (Other); Ontario Rheumatology Association (Unknown); Ontario Best Practices Research Initiative (Unknown)
Responsible Party: Principal Investigator, Dr. Mary Bell, Rheumatologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AHRT-2015
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Inflammatory Arthritis
Keywords: Psoriatic arthritis; Ankylosing spondylitis; Rheumatoid arthritis; Seronegative
MeSH Terms: conditions — Arthritis; Arthritis, Psoriatic; Spondylitis, Ankylosing; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapist Triage (Experimental): All subjects in this group will be triaged by an extended role occupational or physical therapist prior to their visit with the rheumatologist.
  Interventions: Other: Therapist Triage

INTERVENTIONS:
Other: Therapist Triage — An extended role occupational or physical therapist will triage each subject in the study to determine the urgency of their case and how soon they need to see the rheumatologist.

SUMMARY:
There is accumulating evidence that early treatment leads to better outcomes for patients with inflammatory arthritis (IA). Triage, which is the process of identifying the urgency of a patient's disease state efficiently and correctly, may facilitate early referral to a rheumatologist. Several studies have suggested that placing allied health professionals (occupational therapists, physical therapists, nurses, etc.) in a triage roll may reduce wait time for patients with suspected IA. The goal of this investigation will be to demonstrate the system-level impact of an Arthritis Society extended role occupational therapist (OT) or physical therapist (PT) working in a triage role in improving access to rheumatologists for people with IA. In this study two groups will be observed: intervention and "usual care" as determined by historical chart review. Wait times will be compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* New referrals from a GP
* Adults with possible IA (determined by rheumatologist through paper triage)

Exclusion Criteria:

* Currently on a disease-modifying antirheumatic drug (DMARD)
* Previously seen by a rheumatologist.
* FM, non-IA OA; soft tissue rheumatism; mechanical LBP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to first visit with the rheumatologist (wait time) | 3 months

SECONDARY OUTCOMES:
Time to diagnosis | 3 months
Time to treatment (disease-modifying antirheumatic drug) | 3 months